CLINICAL TRIAL: NCT01049672
Title: An Open-label Pilot Comparison Between Alfentanil and Diamorphine for Palliative Care Patients Who Require Subcutaneous Opioids
Brief Title: Diamorphine or Alfentanil for Subcutaneous Use in Hospice In-patients?
Acronym: DASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gloucestershire Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Paul Perkins, Chief Investigator, Gloucestershire Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 07/Q0104/47
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Alfentanil; Heroin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alfentanil (Active Comparator): Hospice in-patients who require subcutaneous strong opioid administration will be given alfentanil
  Interventions: Drug: Alfentanil
- Diamorphine (Active Comparator): Hospice in-patients who require strong opioids will be given diamorphine
  Interventions: Drug: Diamorphine

INTERVENTIONS:
Drug: Alfentanil — Titrated to a maximum dose of 50mg in 24 hours subcutaneously
  Arms: Alfentanil
Drug: Diamorphine — Titrated to a maximum dose of 500mg in 24 hours given subcutaneously
  Arms: Diamorphine

SUMMARY:
OBJECTIVES:

How does Alfentanil compare with the standard drug Diamorphine for subcutaneous analgesia in the palliative care setting?

STUDY DESIGN:

An open-label pilot comparison between alfentanil and diamorphine for palliative care patients who require subcutaneous opioids.

DETAILED DESCRIPTION:
STUDY DESIGN

Study 1 - Open Label Pilot Day - 1 Hospice in-patients who are thought by a clinician to need subcutaneous strong opioids will be asked if they wish to take part in the study.

They will be given a patient information leaflet and a 'cooling off period' (a minimum of 1 day) to think about it. If the clinician feels that strong parenteral opioids are needed diamorphine will be commenced immediately (as standard practice).

Day 0 If the patient agrees to take part in the trial they will be asked to complete a consent form and this will be stored with the patient's notes.

The following assessments will be performed:

1. McGill Pain Questionnaire Short Form(MPQ-SF)
2. Brief Pain Inventory Short Form (BPI-SF)These measures were recommended by an EAPC Expert Working Group for pain syndrome characterization
3. Memorial Delirium Assessment Scale (MDAS). This has been validated in an advanced cancer population and used recently with hospice in-patients.
4. Nausea Visual Analogue Scale (VAS)
5. Nausea Duration over last 24 hours
6. Number of vomits in previous 24 hours

Randomisation Once baseline measures are completed the participant will be randomised using the next available of a series of numbered, opaque, sealed envelopes. These will be prepared remotely. Blocking will be used to prevent an imbalance in terms of the number allocated to each group. Block size will be appropriate to the size of the study and not be divulged to the investigators responsible for consent and revealing the allocation. This will reduce the risk of investigators anticipating the allocation for particular patients. A study log will be kept on site where participant details will be completed before the envelope is opened.

Subsequent Days

On each subsequent day the following assessments will be performed:

1. BPI-SF
2. MDAS
3. Nausea VAS
4. Number of vomits in previous 24 hours

   In addition the following measurements will be taken:
5. Stool chart for previous 24 hours
6. Breakthrough medication (number of doses and dosage) used
7. Laxatives taken
8. Other changes to medication

Patients will cease participation after assessment on day 7.

ELIGIBILITY:
Inclusion Criteria:

1. To be thought by a hospice doctor to require parenteral strong opioids.
2. To have an estimated prognosis of less than 1 year.

Exclusion Criteria:

1. Inability to read English sufficiently to be able to complete assessment questionnaires.
2. Confusion sufficient so that patient is unable to complete questionnaires.
3. Weakness or fatigue sufficient so that patient is unable to complete questionnaires.
4. Radiotherapy to source of pain in last 4 weeks.
5. Change in corticosteroid dose in last week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
The change in MDAS will be calculated from day 0 to day 3 and compared between the two groups using a t-test if the data are sufficiently normally distributed, or the Mann-Whitney U test otherwise. | day 3

SECONDARY OUTCOMES:
Change in MDAS between Days 0 and 7 | Day 7
  The change in MDAS will be calculated from day 0 to day 7 and compared between the two groups using a t-test if the data are sufficiently normally distributed, or the Mann-Whitney U test otherwise.
The change in the BPI-SF | Day 3
  The change in BPI-SF will be calculated from day 0 to day 3 and compared between the two groups using a t-test if the data are sufficiently normally distributed, or the Mann-Whitney U test otherwise.
The change in BPI-SF | Day 7
  The change in BPI-SF will be calculated from day 0 to day 7 and compared between the two groups using a t-test if the data are sufficiently normally distributed, or the Mann-Whitney U test otherwise.
The difference in proportion of patients taking laxatives | Day 7
  The difference in proportion of patients taking laxatives will be compared between the two groups using the confidence interval on the difference of two proportions.
The change in nausea visual analogue scale | Day 3
  The change in nausea visual analogue scale will be calculated from day 0 to day 3 and compared between the two groups using a t-test if the data are sufficiently normally distributed, or the Mann-Whitney U test otherwise.
Change in the number of vomits | Day3
  The change in number of vomits will be calculated from day 0 to day 3 and compared between the two groups using a t-test if the data are sufficiently normally distributed, or the Mann-Whitney U test otherwise.
Change in nausea visual analogue scale | Day 7
  The change in nausea visual analogue scale will be calculated from day 0 to day 7 and compared betwen the two groups using a t-test if the data are sufficiently normally distributed, or the Mann-WhitneyU test otherwise
Change in the number of vomits | Day 7
  The change in number of vomits will be calculated from day 0 to day 7 and compared betwen the two groups using a t-test if the data are sufficiently normally distributed, or the Mann-Whitney U test otherwise.
Change in the total dosage of breakthrough medication (number of doses x dosage) | Day 3
  The change in the total dosage of breakthrough medication will be calculated from day 0 to day 3 and compared betwen the two groups using a t-test if the data are sufficiently normally distributed, or the Mann-WhitneyU test otherwise
Change in the total dosage of breakthrough medication (number of doses x dosage) | Day 7
  The change in the total dosage of breakthrough medication will be calculated from day 0 to day 7 and compared betwen the two groups using a t-test if the data are sufficiently normally distributed, or the Mann-WhitneyU test otherwise

CONTACTS AND LOCATIONS:
Overall Officials: Paul Perkins, MBBCh FRCP, Principal Investigator — Gloucestershire Hospitals NHS Foundation Trust
Locations (1):
- Sue Ryder Care Leckhampton Court Hospice, Cheltenham, Gloucestershire, United Kingdom